CLINICAL TRIAL: NCT05882656
Title: Quality of Life, Functional Outcomes and Costs in Patients Undergoing Primary Total Hip Arthroplasty
Brief Title: Quality of Life, Functional Outcomes and Costs in Hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 03.006.P.35.1
Record Dates: First submitted 2023-05-11; First posted 2023-05-31 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-05

CONDITIONS: Hip Arthropathy
Keywords: hip arthroplasty; hip replacement; quality of life; functional outcomes; costs; cost-utility analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hip arthroplasty: All adult patients undergoing primary total hip replacement surgery at the Traumatology, Orthopedics and Joint Pathology Clinic of the I.M. Sechenov First Moscow State Medical University (Sechenov University) who meet the inclusion criteria (described below) will be included.
  Interventions: Other: Questionnaire administration

INTERVENTIONS:
Other: Questionnaire administration — All study participants will be surveyed with the EQ-5D-5L questionnaire to measure their quality of life indicators before the primary total hip arthroplasty and after the surgery (on 4 dates over a 1-year period); the WOMAC questionnaire to measure their functional outcomes before the primary total hip arthroplasty and after the surgery (on 4 dates over a 1-year period); the costs questionnaire to measure direct and indirect costs borne by patients because of their condition before the primary total hip arthroplasty and after the surgery (on 4 dates over a 1-year period).

SUMMARY:
This prospective observational study aims to collect and analyse data on functional outcomes, quality of life indicators, and costs in patients undergoing primary total hip arthroplasty (hip replacement) surgery.

DETAILED DESCRIPTION:
Primary total hip replacement surgery (also called primary total hip arthroplasty) has been shown to be a safe and reliable procedure for the treatment of degenerative joint disease, which can improve the functional and overall quality of life among patients. This prospective observational study aims to explore how undergoing these surgeries affects patients' functional outcomes and quality of life indicators. Another purpose of this research is to evaluate the costs that generate from this surgical intervention and relate them to the gains in functional outcomes and quality of life measures by conducting cost-utility analysis (CUA).

Participants of this study will be men and non-pregnant women over the age of 18 who are undergoing primary total hip replacement surgery at the Traumatology, Orthopedics and Joint Pathology Clinic of the I.M. Sechenov First Moscow State Medical University (Sechenov University). At this facility, around 300 total hip replacement surgeries are performed annually.

Functional outcomes and quality of life indicators will be measured with validated questionnaires. The Western Ontario and McMaster Universities Arthritis Index (WOMAC) will be used to measure functional outcomes in patients undergoing hip arthroplasty, the 5-level version of the EuroQol-5 Dimension questionnaire (EQ-5D-5L) will be used to measure their health-related quality of life. Questionnaires will be administered to patients before they undergo the procedure and on several follow-up dates (6 weeks, 3 months, 6 months, 1 year after the procedure). Before the surgery the questionnaires will be provided to patients in print form. At other points in time the questionnaires will be administered over the phone or via online forms (way of questionnaire administration depends on the choices of patients).

In addition to tracking changes in patients' functional outcomes and quality of life indicators, patients will be surveyed about all direct and indirect costs generated from seeking treatment for their condition, undergoing the replacement surgery, and the rehabilitation process. A small sample of patients will be interviewed about the costs borne by them to produce a questionnaire which will be used to survey the other patients. Cost information will be collected at the same points in time and in the same formats as stated above (printed questionnaires, telephone surveys, online forms). Financial data for calculating costs borne by the clinic will be obtained from the cost accounting system of the facility after each patient's discharge. Afterwards, the collected cost information will be applied to the CUA. Using quality-adjusted life-years (QALYs) and monetary estimates of costs, Average Cost-Utility Ratios (ACURs) will be calculated for primary total hip replacement surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged 18 years and over
* Patient is willing and able to provide written informed consent to participate in the study including the pre-surgery questionnaire and all post-surgical follow-up questionnaires
* Patients is diagnosed with degenerative joint disease and are admitted to the Traumatology, Orthopedics and Joint Pathology Clinic of the I.M. Sechenov First Moscow State Medical University (Sechenov University) to undergo primary total hip arthroplasty

Exclusion Criteria:

* Patient is unable to provide written consent due to illness or personal circumstances
* Patient is cognitively unable to complete study questionnaires
* Patient refuses to participate in any of the pre-surgery and post-surgical outcome measures (e.g., refuses to provide their contact information for follow-up surveys)
* Patient has an existing condition that would compromise their participation and follow-up in the study (e.g., neuromuscular and psychiatric disorders, musculoskeletal cancer)
* Patient is a pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with degenerative joint disease who are undergoing primary total hip arthroplasty at the Traumatology, Orthopedics and Joint Pathology Clinic of the I.M. Sechenov First Moscow State Medical University (Sechenov University)
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in cost-utility of the primary total hip arthroplasty | Baseline (before surgery), 6 weeks after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  As part of the cost-utility analysis (CUA), the Average Cost-Utility Ratio (ACUR) will be calculated for each time frame after the surgery. ACUR is equal to average health-related costs generated over a time frame divided by average Quality-Adjusted Life years (QALYs) gained over the same time frame. Health-related costs will include all direct and indirect costs before and after surgery (from questionnaires administered to patients and financial data taken from the cost accounting system of the facility). Data on health-related quality of life collected using the EuroQol-5 Dimension questionnaire (EQ-5D-5L) will inform the QALYs calculation.
Change in functional outcomes measured by total scores of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) questionnaire | Baseline (before surgery), 6 weeks after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  The WOMAC questionnaire consists of 24 questions. The overall WOMAC score (index) is determined by summing the scores across the three dimensions of pain (score ranges from 0 to 20), stiffness (score ranges from 0 to 8), and physical function (score ranges from 0 to 68).
Change in quality of life indicators measured by the 5-level version of the EuroQol-5 Dimension questionnaire (EQ-5D-5L) health profile (state), index and the visual analogue scale score (EQ VAS) | Baseline (before surgery), 6 weeks after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  The EQ-5D-5L questionnaire consists of 5 questions in 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In the 5-level version of the questionnaire, each domain has 5 levels. The 5 answers to the 5 questions are combined into a 5-digit number that describes the patients' health profile (state). The 5-digit number can be converted into a single summary index value, which reflects how good or bad a person's health is relative to the general population of a country or region. Another part of the questionnaire is the EQ-VAS which records the patients' self rated-health on a scale from 0 to 100, where 0 = the worst imaginable health and 100 = the best imaginable health.

SECONDARY OUTCOMES:
Level of patients' satisfaction with the primary total hip arthroplasty procedure and overall treatment at the facility | Up to 7 days after the surgery
  This outcome measure consists of patients' answers to two questions:
  * Patients will be asked to rate their level of satisfaction with the surgery, treatment provided at the clinic and their overall experience at the facility on a 0-10 numeric rating scale, where 0 = lowest level of satisfaction and 10 = highest level of satisfaction.
  * Patients will be asked whether they would choose to undergo this surgery at the same facility again if they had to (yes/no question).

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Aleksandrova, Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- Traumatology, Orthopedics and Joint Pathology Clinic of the I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No